CLINICAL TRIAL: NCT02751216
Title: EEG Mapping During High Frequency/High Density Spinal Cord Stimulation in Patients With Failed Back Surgery Syndrome
Acronym: EEGInspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, Prof. dr., Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EEGInspiration1
Record Dates: First submitted 2016-04-18; First posted 2016-04-26 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Failed Back Surgery Syndrome
Keywords: high frequency / high density spinal cord stimulation; EEG; conditioned pain modulation
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spinal cord stimulation (Experimental)
  Interventions: Other: EEG recording + pain protocol

INTERVENTIONS:
Other: EEG recording + pain protocol

SUMMARY:
This study is an interventional, observatory single center trial investigating the functional connectivity of the electrical brain activity in high frequency/high density spinal cord stimulation in failed back surgery syndrome patients with back and leg pain.

DETAILED DESCRIPTION:
Based on the reimbursement rules in Belgium, a trial implantation of 4 weeks is necessary before implanting the definitive neurostimulator. The definitive neurostimulator will be implanted minimum 4 weeks after the trial implantation, when the patient reports more than 50% pain reduction and/or more than 50% reduction in pain medication.

Patients who are included in this study will have four extra study visits at the University Hospital Brussels. The first assessment will take place during the week prior to surgery, the second minimal one month after definitive implantation of the stimulator. The assessments consist of filling in the Pittsburgh Sleep Quality Index (PSQI) and the Pain Catastrophizing Scale (PCS) and recording brain activity before and during the pain protocol. Additionally, patients will wear an Actiwatch for measuring sleep patterns and fill in a VAS diary (back and leg pain separately), one month before the baseline assessment and one month before the second assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old.
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Diagnosis of FBSS with predominant leg pain (VAS) > 5) and non-dominant back pain.
4. Cognitive and language functioning enabling coherent communication between the examiner and the subject;
5. Failed conservative treatments for pain including but not limited to pharmacological therapy and physical therapy
6. Stable neurologic function in the past 30 days
7. In the opinion of the Investigator, the subject is psychologically appropriate for the implantation for an active implantable medical device
8. Subject is able to provide written informed consent
9. Subject speaks Dutch or French.

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing, or plans to become pregnant during the course of the trial
2. Subject has had radiofrequency treatment of an intended target DRG within the past 3 months
3. Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator, deep brain stimulator or intrathecal drug pump
4. Subject is unable to operate the device or has no relative available.
5. Subjects with indwelling devices that may pose an increased risk of infection
6. Subjects currently has an active infection
7. Subject has, in the opinion of the Investigator, a medical comorbidity that contraindicates placement of an active medical device
8. Subject has participated in another clinical investigation within 30 days
9. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
10. Subject has been diagnosed with cancer in the past 2 years
11. Life expectancy < 6 months
12. Imaging (MRI, CT, x-ray) findings within the last 12 months that, in the Investigator's opinion, contraindicates lead placement
13. Existing extreme fear for entering MRI
14. General contraindication for MRI (pacemaker, etc…)
15. Age male/female patient <18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Functional connectivity | The change between baseline and 1 month after definitive implantation of the neurostimulator
  EEG recordings to measure functional connectivity in the brain

SECONDARY OUTCOMES:
Functioning of the descending inhibitory pathway | The change between baseline and 1 month after definitive implantation of the neurostimulator
  Functioning of the descending pathway will be measured with the conditioned pain modulation paradigm by using electrical stimulation and cold water
Visual Analogue Scale (VAS) pain diary | Three times every day (morning, afternoon and evening), starting 1 month before baseline measurements up to the second measurement 1 month after definitive implantation of the neurostimulator (at study completion).
Objective sleep quality will be measured using the Actiwatch spectrum plus (Respironics). | The difference between 1 month before baseline measurements and 1 month before the second measurement (1 month after definitive implantation).
  This compact and lightweight electronic device similar in size to a wristwatch is worn on the non-dominant hand, and measures and records sleep quality
Pain Catastrophizing | The change between baseline and 1 month after definitive implantation of the neurostimulator
  Pain catastrophizing is assess be using the 'pain catastrophizing scale'.
Subjective sleep quality | The change between baseline and 1 month after definitive implantation of the neurostimulator
  Subjective sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI).

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Moens, Prof. dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Vlaams Brabant, Belgium

REFERENCES:
- [Background] De Ridder D, Vanneste S. Burst and Tonic Spinal Cord Stimulation: Different and Common Brain Mechanisms. Neuromodulation. 2016 Jan;19(1):47-59. doi: 10.1111/ner.12368. Epub 2015 Nov 20. PMID 26586145
- [Background] Moens M, Marien P, Brouns R, Poelaert J, De Smedt A, Buyl R, Droogmans S, Van Schuerbeek P, Sunaert S, Nuttin B. Spinal cord stimulation modulates cerebral neurobiology: a proton magnetic resonance spectroscopy study. Neuroradiology. 2013 Aug;55(8):1039-1047. doi: 10.1007/s00234-013-1200-7. Epub 2013 May 12. PMID 23665999
- [Derived] Goudman L, Brouns R, De Groote S, De Jaeger M, Huysmans E, Forget P, Moens M. Association Between Spinal Cord Stimulation and Top-Down Nociceptive Inhibition in People With Failed Back Surgery Syndrome: A Cohort Study. Phys Ther. 2019 Jul 1;99(7):915-923. doi: 10.1093/ptj/pzz051. PMID 30916768